CLINICAL TRIAL: NCT02595684
Title: Effect of Tadalafil on Insulin Secretion and Insulin Sensitivity in Obese Men.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Senior Researcher, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TADALAFIL-OB
Record Dates: First submitted 2015-09-09; First posted 2015-11-03 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: Obesity; Tadalfil; Insulin secretion; Insulin sensitivity
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tadalafil (Experimental): Tadalafil capsules
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Calcined magnesia capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil capsules: 5 mg, one per day, at night, during 28 days.
  Other Names: Tadalafilo
  Arms: Tadalafil
Drug: Placebo — Calcined magnesia capsules: one per day, at night, during 28 days.
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
Obesity is a chronic disease of multifactorial etiology that develops from the interaction of the influence of nutritive , metabolic , cellular and molecular psychological factors.

Tadalafil is Is a drug inhibiting the enzyme phosphodiesterase-5 (PDE-5), responsible for inactivating the vasodilator nitric oxide. USING paragraph was mainly treat erectile dysfunction, and recently approved for the treatment of pulmonary hypertension , it is innovative because of its longer life means, provides efficacy after 36 hours and the highest selectivity.

The aim of this study is to evaluate the effect of tadalafil on insulin sensitivity and insulin secretion in obese men.

The investigators hypothesis is that the administration of tadalafil improve the insulin sensitivity and insulin secretion in obese men.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial in 18 men aged between 30 and 50 years with obesity (BMI 30-39.9) according to the World Health Organization (WHO) criteria without treatment.

They will be assigned randomly in two groups of 9 patients, each to receive 5 mg of tadalafil or placebo every day at night during 28 days.

There will be evaluated Insulin secretion, both first phase of insulin secretion by Stumvoll Inex as well as Total Insulin Secretion by Area Under the Curve of glucose and insulin and Insulinogenic Index, and Insulin sensitivity by Matsuda index.

Waist circumference, glucose and insulin levels, lipid profile and blood pressure are going to be load will be evaluated before and after intervention in both groups.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2, will be used for differences inter-group Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. Will be considered statistical significance p ≤0.05.

This protocol was approved by a local Ethics Committee and written informed consent will be obtained from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age: 30-50 years
* BMI: 30 to 39.9 kg/m²
* No Pharmacotherapy during the last 3 months
* Signature Consent under Information

Exclusion Criteria:

* Cholesterol: ≥ 240 mg / dl
* Triglycerides: ≥ 400 mg / dl
* Fasting glucose: ≥ 126 mg / dl
* Diabetes mellitus.
* Hypertension
* Patients with renal, liver and / or thyroid disease
* Consumption of drugs with known effects on glucose or insulin metabolism.
* Use of cigar and / or drugs
* Hypersensitivity to tadalafil

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel González-Ortíz, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapéutica Experimental y Clínica, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (7.9) | 38.4 (6.4) | 39.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Mexico | 9 | 9 | 18
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 4.9 (0.4) | 4.8 (0.7) | 4.85 (0.55)
Postprandial Glucose [Mean (Standard Deviation); unit: mmol/L] | 6.6 (1.9) | 5.4 (1.3) | 6 (1.6)
First Phase of Insulin [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
  index | 1332 (487) | 1135 (598) | 1233.5 (542.5)
Total Insulin Secretion [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion
  index | 0.82 (0.45) | 0.45 (0.21) | 0.64 (0.33)
Insulin Sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 4.6 (1.2) | 5.0 (2.9) | 4.8 (2.05)
Body Weight [Mean (Standard Deviation); unit: kg] | 98.2 (14.4) | 98.9 (10.4) | 98.55 (12.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (3.3) | 33.3 (3.7) | 33.35 (3.5)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 111 (9) | 110 (13) | 110.5 (11)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.9 (1.0) | 1.9 (0.9) | 1.9 (0.95)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.6 (1.2) | 4.5 (0.8) | 4.55 (1.0)
High Density LIpoprotein cholesterol (HDL-c) [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.3) | 1.0 (0.2) | 1.05 (0.25)
Low density lipoprotein cholesterol (LDL-c) [Mean (Standard Deviation); unit: mmol/L] | 2.7 (0.7) | 2.6 (0.5) | 2.65 (0.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 120 (8) | 120 (10) | 120 (9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81 (7) | 76 (8) | 78.5 (7.5)
Body Fat [Mean (Standard Deviation); unit: %] | 33.3 (6.6) | 31.0 (2.8) | 32.1 (4.8)
Area under the curve (AUC) glucose [Mean (Standard Deviation); unit: mmol*h/L] — The area under the curve (AUC) of glucose, (0.5 * glucose (G) 0´ + (G 30´+G 60´ + G 90´) + 0.5 * G 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperglycemia.
  mmol*h/L | 508 (87) | 513 (146) | 511 (117)
Area under the curve (AUC) insulin [Mean (Standard Deviation); unit: pmol*h/L] — The area under the curve (AUC) of insulin, (0.5 * Insulin (I) 0´ + (I 30´+I 60´ + I 90´) + 0.5 * I 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperinsulinemia.
  pmol*h/L | 285 (114) | 326 (181) | 307 (146)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose
Description: Fasting glucose will be evaluated at baseline and Day 28 with enzymatic-colorimetric.
Time Frame: Fasting glucose at Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol/L | 4.8 (0.6) | 5.0 (0.5)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.327, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.635, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Postprandial Glucose
Description: Postprandial glucose will be evaluated at baseline and Day 28 after a oral glucose. tolerance test with enzymatic-colorimetric techniques.
Time Frame: Postprandial glucose at Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol/L | 6.3 (2.1) | 6.5 (2.3)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.380, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.441, Wilcoxon (Mann-Whitney)

3. Primary Outcome: First Phase of Insulin Secretion
Description: First phase of insulin secretion will be calculated at baseline and Day 28 with Stumvoll Index.
  Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
Time Frame: First phase of insulin secretion at Day 28
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
index | 1602 (800) | 1194 (490)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0515, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.953, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Total Insulin Secretion
Description: Total insulin secretion will be calculated at baseline and Day 28 with Insulinogenic Index.
  The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔAUC insulin/ΔAUC glucose), the entered values reflect the total insulin secretion
Time Frame: Total insulin secretion at Day 28
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
index | 0.52 (0.29) | 0.61 (0.27)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.314, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.594, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity will be calculated at baseline and Day 28 with Matsuda Index.
  Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
Time Frame: Insulin sensitivity at Day 28
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
index | 4.8 (3.1) | 4.9 (2.5)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.767, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.779, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Area Under the Curve (AUC) Glucose
Description: Area under the curve of glucose measured at baseline and Day 28. The area under the curve (AUC) of glucose, (0.5 * glucose (G) 0´ + (G 30´+G 60´ + G 90´) + 0.5 * G 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperglycemia.
Time Frame: AUC at Day 28
Measure: Mean (Standard Deviation); unit: mmol*h/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol*h/L | 503 (137) | 522 (135)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.859, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.767, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Area Under the Curve (AUC) Insulin
Description: Area under the curve of insulin measured at baseline and Day 28. The Area Under the Curve (AUC) of insulin, (0.5 * Insulin (I) 0´ + (I 30´+I 60´ + I 90´) + 0.5 * I 120´) * 30; has been widely used for calculating the glycemic index and for evaluating the efficacy of medications for postprandial hyperinsulinemia.
Time Frame: AUC at Day 28
Measure: Mean (Standard Deviation); unit: pmol*h/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
pmol*h/L | 291 (160) | 262 (110)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.374, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.953, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Body Weight
Description: The body weight will be measured at baseline and Day 28 by Electrical bioimpedance.
Time Frame: Body Weight at Day 28
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
kg | 99.1 (14.4) | 98.2 (9.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.594, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.085, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Body Mass Index
Description: The Body Mass Index will be measured at baseline and Day 28 by Quetelet Index Formula.
Time Frame: Body Mass Index at Day 28
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
kg/m^2 | 33.7 (3.3) | 33.1 (3.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.594, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.086, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Waist Circumference
Description: Waist circumference was evaluated at baseline and at Day 28 with a flexible tape.
Time Frame: Waist circumference at Day 28
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
cm | 112 (9) | 112 (13)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.285, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.854, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Triglycerides
Description: Triglycerides levels will be evaluated at baseline and Day 28 with enzymatic-colorimetric techniques.
Time Frame: Triglycerides levels at Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol/L | 2.3 (1.9) | 2.4 (2.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.374, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.263, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Total Cholesterol
Description: Total cholesterol levels will be evaluated at baseline and Day 28 with enzymatic-colorimetric techniques.
Time Frame: Total cholesterol levels at Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol/L | 4.4 (0.9) | 4.3 (1.3)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.859, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.374, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL-c)
Description: High density lipoprotein cholesterol (HDL-c) levels will be evaluated at baseline and Day 28 with enzymatic-colorimetric techniques.
Time Frame: HDL-c levels at Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol/L | 1.1 (0.2) | 1.1 (0.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.722, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.953, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Low Density Lipoprotein Cholesterol (LDL-c)
Description: Low density lipoprotein cholesterol (LDL-c) levels will be evaluated at baseline and Day 28 with Friedewald formula.
Time Frame: LDL-c levels at Day 28
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmol/L | 2.3 (0.5) | 2.2 (0.8)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.260, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.314, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Systolic Blood Pressure
Description: The systolic blood pressure was evaluated at baseline and Day 28 with a digital sphygmomanometer.
Time Frame: Systolic Blood Pressure at Day 28
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmHg | 120 (6) | 115 (8)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.058, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.952, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Diastolic Blood Pressure
Time Frame: Diastolic Blood Pressure at Day 28
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
mmHg | 77 (6) | 73 (7)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.128, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.108, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Body Fat
Description: The body fat will be measured at baseline and Day 28 by Electrical bioimpedance in %
Time Frame: Body fat at Day 28
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 9 | 9
percentage of fat | 33.7 (3.3) | 33.1 (3.7)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.092, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tadalafil; Test type: Superiority; p = 0.374, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Throughout the study, an average of 28 days
Arm/Group | Tadalafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/9 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=9) | Placebo (N=9)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Chills (Infections and infestations) | 1 (1) | 0 (0)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Edema (Renal and urinary disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes